CLINICAL TRIAL: NCT02596711
Title: Project Impact 2: A Culturally Tailored Smoking Cessation Intervention for Latino Smokers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0585; K01CA160670 (NIH); NCI-2016-00193 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Tobacco Use Cessation; Cancer Prevention
Keywords: Cancer Prevention; Tobacco Use Cessation; Nicotine Patch; NRT; Questionnaires; Surveys; Carbon Monoxide Test; CO; Health Education; Handouts; Pamphlets; Counseling sessions
MeSH Terms: conditions — Tobacco Use Cessation; Health Education | interventions — Tobacco Use Cessation Devices; Surveys and Questionnaires; Carbon Monoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Health Education (HE) Group (Experimental): Participants receive general health education and handouts. Participants attend 3 counseling sessions during the study. Each of these counseling sessions are audio recorded. Counselor discusses a health topic (such as sleep, nutrition, and exercise) and how it relates to participant and their smoking. Participants receive 12 weeks of Nicotine Replacement Therapy (NRT).
  Interventions: Drug: Nicotine Patch; Behavioral: Questionnaires; Other: Carbon Monoxide (CO) Test; Behavioral: Health Education and Handouts; Behavioral: Counseling Sessions
- Culturally Tailored Smoking Cessation (CTSC) Group (Experimental): Participants given reading materials that highlight how aspects of their culture relate to health, smoking and quitting. Participants attend 3 counseling sessions during the study. Each of these counseling sessions are audio recorded. Participant and counselor discuss how smoking and their culture may relate to each other. Participants receive 12 weeks of Nicotine Replacement Therapy (NRT).
  Interventions: Drug: Nicotine Patch; Behavioral: Questionnaires; Other: Carbon Monoxide (CO) Test; Behavioral: Culturally Tailored Reading Materials; Behavioral: Counseling Sessions
- Culturally Tailored Smoking + Adherence Enhancement (AE) Group (Experimental): Participants given reading materials that highlight how aspects of their culture relate to health, smoking and quitting. Participants attend 3 counseling sessions during the study. Each of these counseling sessions are audio recorded. Participants receive additional talks related to smoking cessation tailored to their culture. Participants receive 12 weeks of Nicotine Replacement Therapy (NRT).
  Interventions: Drug: Nicotine Patch; Behavioral: Questionnaires; Other: Carbon Monoxide (CO) Test; Behavioral: Culturally Tailored Reading Materials; Behavioral: Counseling Sessions

INTERVENTIONS:
Drug: Nicotine Patch — Participants receive 4 weeks of 21 mg, 4 weeks of 14 mg, and 4 weeks of 7 mg patches.
  Other Names: NRT
Behavioral: Questionnaires — Questionnaires regarding tobacco and alcohol use, culture, religion, and sense of control completed at baseline, at weeks 2 and 6, and at 3 and 6 months after baseline.
  Other Names: Surveys
Other: Carbon Monoxide (CO) Test — Carbon monoxide (CO) test given at baseline, at weeks 2 and 6, and at 3 and 6 months after baseline.
Behavioral: Health Education and Handouts — Participants receive general health education and handouts.
  Other Names: Pamphlets
  Arms: Health Education (HE) Group
Behavioral: Culturally Tailored Reading Materials — Participants given reading materials that highlight how aspects of their culture relate to health, smoking and quitting.
  Other Names: Pamphlets
  Arms: Culturally Tailored Smoking + Adherence Enhancement (AE) Group; Culturally Tailored Smoking Cessation (CTSC) Group
Behavioral: Counseling Sessions — Participants attend 3 counseling sessions during the study.

SUMMARY:
The goal of this research study is to learn how 3 different kinds of counseling treatments may help individuals to quit smoking.

DETAILED DESCRIPTION:
Baseline Visit:

If you agree to take part in this study, the following tests and procedures will be performed at the beginning of the study:

* You will complete 10 questionnaires about your demographics (age, race, sex, and so on), medical history, smoking status, alcohol use, religion, how "in control" you feel of your own life, and cultural background. These should take about 1½ hours to complete.
* You will complete a carbon monoxide (CO) test to measure the level of carbon monoxide in your body. This test involves blowing your breath through a hand-held device.
* You will learn how to keep a diary about your progress in your attempts to quit smoking. °You must bring this diary with you to every visit.
* You will be asked if you have smoked any non-tobacco substances in the last 2 days. If you have, you will provide an additional CO sample 2 days after the last time you smoked the substance.
* If you can become pregnant, you will have a urine pregnancy test. To take part in this study, you must not be pregnant.3
* The total length of the baseline visit will be approximately 2.5 hours.

Study Groups:

You will be randomly assigned (as in the roll of dice) into 1 of 3 study groups. You will have an equal chance of being in each group. This is done because no one knows if one study group is better, the same, or worse than the other group.

Counseling Sessions:

The study group that you are in will determine the way that health information is presented to you in one-on-one counseling sessions.

* If you are in Group 1, you will receive general health education. The counselor will discuss a health topic (such as sleep, nutrition, and exercise) and how it relates to you and your smoking. The counselor will also give you handouts about the health topic.
* If you are in Group 2, you and the counselor will discuss how your smoking and your culture may relate to each other. The counselor will also provide you with reading materials that highlight how aspects of your culture relate to health, smoking and quitting.
* If you are in Group 3, you will receive the same cultural counseling and handouts that Group 2 received. Also, you will have additional talks about the use of drugs to help you stop smoking and some common feelings that Latinos may experience with being unsuccessful when trying to quit. The counselor will also offer you a plan for using medication successfully.

All participants will attend 3 counseling sessions during the study. Each of these counseling sessions will be audio recorded. Your first counseling session will be at baseline. The other two counseling sessions will be at your Week 2 and Week 6 visits (described below).

All participants will be given a 12 week supply of nicotine patches and information about how to use the nicotine patch. At each study visit, you will be given the amount of patches that you need to last you to your next visit, plus a few extra in the event that a patch falls off or is damaged.

During your first counseling session, you will be asked to choose a quit date. This is simply a date that you would like to begin using the patch and make an attempt to not smoke.

Week 2 and Week 6 Study Visits:

At each of these study visits, all participants will have the following procedures:

* You will complete a brief interview about your progress and any side effects you may be having. This should take about 10 minutes to complete.
* You will complete 2 questionnaires about your tobacco use and satisfaction with the study. These should take about 10 minutes to complete.
* You will complete a CO test.
* You will be asked if you have smoked any other substances, such as marijuana, in the last 2 days. If you have, you will provide an additional CO sample 2 days after the last time you smoked the substance.

Follow-Up Visits:

About 3 months and 6 months after baseline, you will have a follow-up visit. At each of these visits, the following tests and procedures will be performed:

* You will complete the same set of questionnaires about your tobacco and alcohol use, culture, religion, and sense of control that you did at your baseline visit.
* You will complete a CO test.
* You will be asked if you have smoked any non-tobacco substances in the last 2 days. If you have, you will provide an additional CO sample 2 days after the last time you smoked the substance.

Length of Study:

Your study participation will be over after you complete the 6-month follow-up visit.

This is an investigational study. Up to 36 people will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 18 years of age
2. Current smoker (>5 cigarettes per day for the past 3 months)
3. Able to speak and read English or Spanish
4. Agree to participate in the study and be available for 6 weeks of treatment and 6 months of follow-up
5. Willing to set a quit date within 2 weeks of enrollment date
6. Identify as being of Latino heritage, ethnicity, or ancestry

Exclusion Criteria:

1. Individuals suffering from any unstable medical condition precluding the use of NRT (Identified using the Medical History Questionnaire given at baseline)
2. Currently using smokeless tobacco, electronic nicotine delivery systems (ENDS), nicotine replacement therapy, or other smoking cessation treatment
3. Pregnant or nursing
4. Suffering from a severe psychiatric disorder (assessed using self-reporting history of psychiatric diagnosis during the phone screening) that would interfere with participation
5. Diagnosis of substance dependence other than nicotine (screened using DSM IV TR criteria) Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition
6. Individuals that do not have access to a working telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcel A. de Dios, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] de Dios MA, Cano MA, Vaughan EL, Childress SD, McNeel MM, Harvey LM, Niaura RS. A pilot randomized trial examining the feasibility and acceptability of a culturally tailored and adherence-enhancing intervention for Latino smokers in the U.S. PLoS One. 2019 Jan 11;14(1):e0210323. doi: 10.1371/journal.pone.0210323. eCollection 2019. PMID 30633744
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Houston metropolitan area (Harris County, Texas) through fliers at community centers and local health clinics as well as through advertisements online and in print newspapers between February of 2016 and January of 2017.
Pre-assignment Details: During baseline visit (prior to randomization), an expired carbon monoxide sample was collected using Bedfont Micro+Smokerlyzer.Additionally, participants able to become pregnant were required to take a routine hCG urine sample pregnancy test to rule out potential pregnancy.An assessment battery was also administered at the baseline visit.
Groups:
- Health Education (HE): Used as the control condition. Participants receive general health education and handouts. Participants attend 3 counseling sessions during the study. Each of these counseling sessions are audio recorded. Counselor discusses a health topic (such as sleep, nutrition, and exercise) and how it relates to participant and their smoking. Participants receive 12 weeks of Nicotine Replacement Therapy (NRT).
- Culturally-Tailored (CT): Participants given reading materials that highlight how aspects of their culture relate to health, smoking and quitting. Participants attend 3 counseling sessions during the study. Each of these counseling sessions are audio recorded. Participant and counselor discuss how smoking and their culture may relate to each other. Participants receive 12 weeks of Nicotine Replacement Therapy (NRT).
- Culturally-Tailored With Adherence Enhancement (CT+AE): Participants given reading materials that highlight how aspects of their culture relate to health, smoking and quitting. Participants attend 3 counseling sessions during the study. Each of these counseling sessions are audio recorded. Participants receive additional talks related to smoking cessation tailored to their culture. Participants receive 12 weeks of Nicotine Replacement Therapy (NRT).
Period: Overall Study
Arm/Group | Health Education (HE) | Culturally-Tailored (CT) | Culturally-Tailored With Adherence Enhancement (CT+AE)
Started | 9 | 8 | 8
Visit 2 | 9 | 7 | 6
Visit 3 | 7 | 8 | 6
3 Month Follow-up | 8 | 6 | 6
6 Month Follow-up | 8 | 6 | 5
Completed | 8 | 6 | 5
Not Completed | 1 | 2 | 3
Not completed — Lost to Follow-up | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Education (HE) | Culturally-Tailored (CT) | Culturally-Tailored With Adherence Enhancement (CT+AE) | Total
Number analyzed (Participants) | 9 | 8 | 8 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 8 | 25
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 45.4 (11) | 46 (10.94) | 40.7 (13.92) | 44.1 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 5 | 5 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 8 | 25
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 2 | 3 | 13
  More than one race | 1 | 2 | 2 | 5
  Unknown or Not Reported | 0 | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 8 | 8 | 25

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility & Acceptability
Description: The central aim of this pilot study was to evaluate the feasibility and acceptability of our treatment interventions. As such, we examined between-group differences on session satisfaction. After completing each session, participants anonymously rated their level of satisfaction with the counseling session. This investigator created scale (Session Satisfaction Scale) used a 5-point Likert scale (from 1 = "Extremely Unsatisfied" to 5 = "Extremely Satisfied"). Mean satisfaction scores were computed for each participant as the average of all session satisfaction scores. Higher scores indicating greater levels of satisfaction. Treatment group session satisfaction group means were tabulated by group (calculated as the average for all participants in each treatment group) and used as a proxy measure of overall intervention acceptability and feasibility.
Time Frame: Averaged across 3 study visits (Week 0 to Week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Health Education (HE) | Culturally-Tailored (CT) | Culturally-Tailored With Adherence Enhancement (CT+AE)
Number analyzed (Participants) | 9 | 8 | 8
score on a scale | 4.87 (0.35) | 4.71 (0.48) | 4.83 (0.4)

2. Primary Outcome: Patch Adherence: Percentage of Days With Patch
Description: Adherence to NRT patch (days of NRT patch use) collected with the Timeline followback interview procedure.
Time Frame: This outcome was collected at each study timepoint and measured the 12 weeks of NRT patch treatment.
Measure: Mean (Standard Deviation); unit: percentage of NRT patch days
Arm/Group | Health Education (HE) | Culturally-Tailored (CT) | Culturally-Tailored With Adherence Enhancement (CT+AE)
Number analyzed (Participants) | 9 | 8 | 8
percentage of NRT patch days | 64.6 (17.7) | 68.6 (13.66) | 81.3 (3.32)

3. Primary Outcome: Number of Abstinent Participants
Description: Rates of biochemically verified 7-day point prevalence smoking abstinence. Collected with the Timeline Follow-back interview procedure and verified with a expired carbon monoxide testing with a Bedfont Smokelyzer monitor.
Time Frame: Collected at the 3- and 6-month follow-up visits
Measure: Count of Participants; unit: Participants
Arm/Group | Health Education (HE) | Culturally-Tailored (CT) | Culturally-Tailored With Adherence Enhancement (CT+AE)
Number analyzed (Participants) | 9 | 8 | 8
Participants
  3-month follow-up | 4 | 2 | 4
  6-month follow-up | 4 | 2 | 3

ADVERSE EVENTS:
Time Frame: End of treatment and 6 month follow-up
Description: MD Anderson requires that all Protocol PIs and their designees report all Serious Adverse Events and Adverse Events (n=4) to the MD Anderson IRB on an ongoing bases using a systematic approach with standardized forms. SAE's and AE's are reported as they occur and during each continuation reports submission.
Arm/Group | Health Education (HE) | Culturally-Tailored (CT) | Culturally-Tailored With Adherence Enhancement (CT+AE)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/9 | 1/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Education (HE) (N=9) | Culturally-Tailored (CT) (N=8) | Culturally-Tailored With Adherence Enhancement (CT+AE) (N=8)
Nausea and changes in appetite, likely related to increase in patch dosage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rapid heart rate and anxiety, likely related to patch use (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disturbances, anxiety, abnormal taste in mouth, trouble concentrating, sad mood. (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mild sleep disturbance and irratbility. (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep disturbance, constipation, skin irritation and lesion at patch site, lower back pain, phlegm i (General disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the limited scope, the study was not fully powered for conclusive hypothesis testing of group differences on variables of interest. The analytic strategy focused on descriptive statistics and estimation rather than formal hypothesis testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02596711/Prot_SAP_000.pdf